CLINICAL TRIAL: NCT05612152
Title: Choose2Quit: Improving Equity in Smoking Cessation for Low Income Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Case Western Reserve University (Other); MetroHealth System, Ohio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RSG-18-137-01-CPPB
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Referral to Quitline (Active Comparator): Patients who indicate they are ready to quit in the next 30 days are offered an electronic referral to the state quitline for tobacco cessation services.
  Interventions: Other: Referral to Quitline
- Choose2Quit (Experimental): Patients who indicate they are ready to quit in the next 30 days are offered an electronic referral to the Choose2Quit tobacco treatment navigator who walks the patient through choices for tobacco cessation counseling, tobacco cessation medications and other supports (e.g. texting, apps) and facilitates placing referrals, orders and providing information.
  Interventions: Other: Choose2Quit

INTERVENTIONS:
Other: Referral to Quitline — An electronic referral to the state quitline is placed. This prompts the quitline to proactively call the patient to enroll in counseling services.
  Arms: Referral to Quitline
Other: Choose2Quit — An electronic referral to the Choose2quit tobacco cessation navigator is placed. This prompts the navigator to call the patient to review options for tobacco cessation counseling, tobacco cessation medications and other supports.
  Arms: Choose2Quit

SUMMARY:
The goal of this study is to evaluate the effectiveness of a tobacco treatment navigator to improve primary care patient engagement in tobacco cessation support. We compare an ask, advise and connect to the quitline approach vs. the novel tobacco treatment navigator approach on the primary outcomes of receipt of tobacco cessation counseling sessions and receipt of tobacco cessation medications.

DETAILED DESCRIPTION:
Our novel intervention, Choose2Quit, builds on our prior successes with the Ask, Advice, Connect study, but now 1) allows personalized choice of counseling modality (phone, text, web, in-person); 2) conveys the value and low/no-cost availability of medications to support quit attempt success and sends providers the patient's request in e-prescription to transmit to patient's pharmacy; 3) assesses patient's need to manage social barriers to quitting by linking them to Unite-US; and 4) uses an initial phone contact from a recognizable local number, will increase the engagement of patients in cessation treatment and in tobacco cessation. This study aims to:

1. Test the effect of a traditional eReferral vs. a Choose2Quit personalized guidance and choice approach on the ability to contact patients, and the proportion of patients that initiate tobacco cessation treatment, use tobacco cessation medications and make quit attempts.
2. Assess the impact of each intervention arm on equitable engagement in tobacco cessation treatment, medication use and quit outcomes across gender, race and age groups.
3. Evaluate intervention experience from the patient perspective.
4. Evaluate the cost to implement, and per engagement in each of the intervention arms.

The study is accomplished using a 2-arm randomized trial. Randomization into the traditional eReferral vs. Choose2Quit intervention arms will occur at the patient level with a 1:1 group assignment. Individuals that are ready to quit in the next 30 days and are interested in being connected with tobacco cessation resources will be randomized. Randomization of eligible patients occurs automatically with an electronic health record algorithm that routes the eReferral to the Quitline (traditional eReferral) or the Choose2Quit intervention. The Ask-Advise-Connect process is exactly the same for medical assistants; medical assistants and patients are blind to group assignment

ELIGIBILITY:
Inclusion Criteria:

* patient care visit to one of the participating primary care clinics during the study period
* reports current tobacco use
* reports interest in quitting tobacco in the next 30 days
* accepts offer of referral to tobacco cessation support

Exclusion Criteria:

* not interested in quitting in next 30 days
* not interested in assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
receipt of tobacco cessation counseling | 4 weeks after referral
  receipt of 1 or more tobacco cessation counseling sessions from referral sources
receipt of tobacco cessation medications | within 4 weeks after referral
  documentation of orders for nicotine replacement therapy, varenicline or bupropion in electronic health record

SECONDARY OUTCOMES:
7-day point prevalence abstinence | 8 weeks after referral
  7-day point prevalence abstinence from tobacco use